CLINICAL TRIAL: NCT00824733
Title: A Phase II Open-label Study of Subcutaneous CPG ODN (PF03512676) in Combination With Trastuzumab in Patients With Metastatic Breast Cancer
Brief Title: Agatolimod and Trastuzumab in Treating Patients With Locally Advanced or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inaccurate patient accrual for trial
Sponsor: Bhuvaneswari Ramaswamy (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Bhuvaneswari Ramaswamy, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-08153; NCI-2011-03157 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; HER2-positive breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I: Treatment (PF03512676 in combination with Trastuzumab) (Experimental): 12 weekly treatments. Week 1-12 patients will receive Trastuzumab 2mg/kg IV(intervenous infusion). Patients who have not been treated wih Trastuzumab within 4 weeks will receive a loading dose of 4 mg/kg on week 1 and PF-03512676-0.16 mg/kg subcutaneous injection.Correlative studies will be drawn on week 1, 2, 6, 12 and 18.
  Interventions: Drug: Trastuzumab; Drug: PF03512676; Other: Correlative Studies

INTERVENTIONS:
Drug: Trastuzumab — IV at 2 mg/kg over 30 minutes on day 1 of each weekly cycle. Patients who have not received trastuzumab for 4 weeks or more will receive a loading dose of 4 mg/kg over 90 minutes day 1 of the first cycle. The dose of trastuzumab will be based on the patient's actual weight at the start of each 4 week treatment cycle.
  Other Names: Herceptin
Drug: PF03512676 — Patients also receive PF03512676 subcutaneously on days 15 and 22 of course 1 and on days 1, 8, 15, and 22 of all subsequent courses.
  Other Names: agatolimod sodium
Other: Correlative Studies — Blood for performing the correlative studies will be drawn on week 1, 2, 6, 12 and 18.

SUMMARY:
RATIONALE: Biological therapies, such as agatolimod, may stimulate the immune system in different ways and stop tumor cells from growing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving agatolimod together with trastuzumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving agatolimod together with trastuzumab works in treating patients with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the progression-free survival of patients with HER2-overexpressing locally advanced or metastatic breast cancer treated with trastuzumab (Herceptin®) and agatolimod sodium.

Secondary

* To determine if agatolimod sodium augments antibody-mediated cytoxicity (ADCC) against trastuzumab-coated target cells by evaluating the ability of patient immune-effector cells to conduct ADCC and produce interferon gamma.

OUTLINE: This is a multicenter study.

Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes on day 1. Patients also receive agatolimod sodium subcutaneously on days 15 and 22 of course 1 and on days 1, 8, 15, and 22 of all subsequent courses. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for correlative laboratory studies. Samples are analyzed for antibody-mediated cytotoxicity (ADCC) by chromium-release assay; IFN-γ production and quantification by flow cytometry and reverse transcriptase-polymerase chain reaction (RT-PCR); and levels of cytokines (IFN-γ and TNF-α) by ELISA.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Locally advanced or metastatic disease
* HER2-overexpressing tumor, defined as 3+ overexpression by IHC and/or HER2 amplified by FISH
* Non-measurable disease allowed
* Achieved partial response, complete response, or stable disease (i.e., no disease progression for ≥ 12 weeks) while on trastuzumab (Herceptin®) and chemotherapy, hormonal therapy alone, or trastuzumab alone

  * Last dose of trastuzumab must have been administered within the past 16 weeks
* No unstable brain metastases

  * Patients with brain metastases are eligible provided they have been stable for ≥ 1 month after surgery or radiotherapy/radiosurgery AND off corticosteroids and anticonvulsants for ≥ 4 weeks
* Hormone receptor status unspecified

PATIENT CHARACTERISTICS:

* ECOG(Eastern Cooperative Oncology Group)performance status (PS) 0-2 (Karnofsky PS 70-100%)
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin > 8 g/dL (transfusion/epoetin alfa allowed)
* Platelet count ≥ 100,000/mm³
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (≤ 5.0 times ULN if known liver metastases)
* Creatinine < 2 mg/mL
* Ejection fraction ≥ 50% by echocardiogram or MUGA
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and for ≥ 3 months after completion of study treatment
* No ongoing or active infection requiring oral or IV antibiotics
* No known autoimmune disorders or antibody-mediated disorders
* No known HIV positivity
* No known history of hepatitis B or C (active and/or previously treated)
* No other malignancies within the past 5 years except nonmelanoma skin cancer or cervical cancer in situ
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 12 weeks since prior chloroquine
* More than 4 weeks since prior growth factors
* More than 4 weeks since prior systemic corticosteroids
* More than 4 weeks since prior chemotherapy, radiotherapy, or monoclonal antibody therapy (except trastuzumab)
* No prior agatolimod sodium
* No prior allogeneic stem cell transplantation
* No prior continuous treatment with single-agent trastuzumab for > 6 months
* No more than 3 prior chemotherapy regimens for metastatic breast cancer
* Any number of prior hormonal therapies allowed
* No other concurrent investigational agents or monoclonal antibodies
* No other concurrent anticancer agents or therapies
* Concurrent bisphosphonates for skeletal metastasis allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-02; Primary Completion 2013-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhuvaneswari Ramaswamy, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I: Treatment (PF03512676 in Combination With Trastuzumab)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I: Treatment (PF03512676 in Combination With Trastuzumab)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: patients]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: PF-03512676 Augments Antibody Mediated Cytoxicity (ADCC)Against Trastuzumab-coated Target Cells in Metastatic HER2 Overexpressing Breast Cancer.
Time Frame: up to 18 weeks
Population: Samples were not analyzed for primary endpoint due to the sample numbers being too small. No data were collected from the samples.
Arm/Group | Arm I: Treatment (PF03512676 in Combination With Trastuzumab)
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-free Survival for Patients With Metastatic Breast Cancer That Are Receiving Trastuzumab Plus PF-03512676
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: up to 18 weeks
Measure: Median (Full Range); unit: weeks
Arm/Group | Arm I: Treatment (PF03512676 in Combination With Trastuzumab)
Number analyzed (Participants) | 6
weeks | 13 [7 to 16]

3. Secondary Outcome: Combination of PF-03512676 and Trastuzumab Induces MIP-1 (Macrophage Inflammatory Protein 1), MCP-1 (Monocyte Chemoattract Protein 1) and RANTES.
Time Frame: up to 18 weeks
Population: The study was terminated early due to poor patient accrual and no data was collected and analyzed.
Arm/Group | Arm I: Treatment (PF03512676 in Combination With Trastuzumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were graded using the NCI Common Toxicity Criteria (CTC) version 3.0.
Arm/Group | Arm I: Treatment (PF03512676 in Combination With Trastuzumab)
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Treatment (PF03512676 in Combination With Trastuzumab) (N=6)
Injection site reaction (General disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Treatment (PF03512676 in Combination With Trastuzumab) (N=6)
fatigue (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Injection site reaction (General disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes